CLINICAL TRIAL: NCT03103880
Title: Assessing the Use of Digital Therapeutic in Adult Asthma Patients: A Remote Observational Study
Brief Title: Assessing the Use of Mobile Technology in Adult Asthma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CoheroHealth (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2017 Observational Study 1.0; NCT05712863 (obsolete NCT alias)
Record Dates: First submitted 2017-03-28; First posted 2017-04-06 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Asthma
Keywords: Patient adherence; Mobile application; Mobile health; Digital therapeutics; Digital health
MeSH Terms: conditions — Asthma; Patient Compliance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- BreatheSmart (Experimental): 104 subjects will be provided with the BreatheSmart platform, which consists of:
  1. HeroTracker sensor that monitors real-time asthma medication adherence
  2. BreatheSmart mobile application that provides patients with real-time alerts, environmental information (weather, pollution, etc.), and the ability to complete questionnaires / surveys.
  Interventions: Device: BreatheSmart

INTERVENTIONS:
Device: BreatheSmart — BreatheSmart is a comprehensive asthma monitoring system that combines a medical device and mobile application that are designed for use with Apple and Android mobile devices. The medical device connects to the mobile application using Bluetooth to facilitate the collection of controlled medication adherence, rescue medication usage, and asthma control.

SUMMARY:
This is a prospective, remote observational study of adults with persistent asthma who are managed on inhaled corticosteroids.

DETAILED DESCRIPTION:
The study consists of one interventional group and all 104 subjects will be included in this group. All subjects will be provided with the HeroTracker package, which includes:

1. HeroTracker sensor that counts dosage and monitors real-time medication adherence
2. BreatheSmart mobile application that sends subjects real-time alerts and allows patients respond to questionnaires / surveys.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide written informed consent
* Male and female adults (aged ≥ 18 years)
* Diagnosis of asthma for at least 6 months
* ICS (inhaled corticosteroid) use for at least 3 months
* Use of a pressurized metered dose inhaler (pMDI) compatible with the HeroTracker
* Possess a compatible smartphone (iOS 8.0 or higher and Android 4.3 or higher)

Exclusion Criteria:

* Currently pregnant or planning to become pregnant during the study period
* Primary language other than English (BreatheSmart mobile app is currently available only in English)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-04-21 (Actual); Primary Completion 2018-08-29 (Actual); Study Completion 2018-08-29 (Actual)

PRIMARY OUTCOMES:
Change in asthma control | 3 months
  Determine change in the asthma control test (ACT), a validated asthma test, in subjects using the BreatheSmart system from baseline to 3 months.
Change in rescue medication usage | 3 months
  Determine change in rescue medication usage in subjects the BreatheSmart system from baseline to 3 months.

SECONDARY OUTCOMES:
Change in controller medication adherence | 3 months
  Obtain medication adherence percentage (that ranges from 0-100%) to asthma inhaled corticosteroids (ICS) at baseline to 3 months.
Acceptability of BreatheSmart system | 3 months
  Acceptability questionnaire (delivered through the BreatheSmart mobile application) that includes subjects' opinion on the platform, features, usability, and usefulness.

CONTACTS AND LOCATIONS:
Overall Officials: Anne Tam, MPH, Study Director — Cohero Health, Inc.
Locations (1):
- Cohero Health, Inc., New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lasmar L, Camargos P, Champs NS, Fonseca MT, Fontes MJ, Ibiapina C, Alvim C, Moura JA. Adherence rate to inhaled corticosteroids and their impact on asthma control. Allergy. 2009 May;64(5):784-9. doi: 10.1111/j.1398-9995.2008.01877.x. Epub 2009 Jan 21. PMID 19183166
- [Background] Chan AH, Harrison J, Black PN, Mitchell EA, Foster JM. Using electronic monitoring devices to measure inhaler adherence: a practical guide for clinicians. J Allergy Clin Immunol Pract. 2015 May-Jun;3(3):335-49.e1-5. doi: 10.1016/j.jaip.2015.01.024. Epub 2015 Apr 1. PMID 25840665
- [Background] Schatz M, Kosinski M, Yarlas AS, Hanlon J, Watson ME, Jhingran P. The minimally important difference of the Asthma Control Test. J Allergy Clin Immunol. 2009 Oct;124(4):719-23.e1. doi: 10.1016/j.jaci.2009.06.053. Epub 2009 Sep 19. PMID 19767070
- [Background] Jia CE, Zhang HP, Lv Y, Liang R, Jiang YQ, Powell H, Fu JJ, Wang L, Gibson PG, Wang G. The Asthma Control Test and Asthma Control Questionnaire for assessing asthma control: Systematic review and meta-analysis. J Allergy Clin Immunol. 2013 Mar;131(3):695-703. doi: 10.1016/j.jaci.2012.08.023. Epub 2012 Oct 8. PMID 23058645
- [Background] Melosini L, Dente FL, Bacci E, Bartoli ML, Cianchetti S, Costa F, Di Franco A, Malagrino L, Novelli F, Vagaggini B, Paggiaro P. Asthma control test (ACT): comparison with clinical, functional, and biological markers of asthma control. J Asthma. 2012 Apr;49(3):317-23. doi: 10.3109/02770903.2012.661008. Epub 2012 Mar 9. PMID 22401649
- [Background] Korn S, Both J, Jung M, Hubner M, Taube C, Buhl R. Prospective evaluation of current asthma control using ACQ and ACT compared with GINA criteria. Ann Allergy Asthma Immunol. 2011 Dec;107(6):474-9. doi: 10.1016/j.anai.2011.09.001. Epub 2011 Oct 5. PMID 22123375
- [Derived] Melvin E, Cushing A, Tam A, Kitada R, Manice M. Assessing the use of BreatheSmart(R) mobile technology in adult patients with asthma: a remote observational study. BMJ Open Respir Res. 2017 Aug 16;4(1):e000204. doi: 10.1136/bmjresp-2017-000204. eCollection 2017. PMID 29071077